CLINICAL TRIAL: NCT00666237
Title: Primary Tube Versus Trabeculectomy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Abbott Medical Optics (Industry); Research to Prevent Blindness (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Steven J. Gedde, Dr, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20071037; EY014801 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma
Keywords: Tube shunt surgery; Trabeculectomy
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants; Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tube shunt surgery group (Experimental): Participants in this group will receive a tube shunt surgery (Baerveldt Glaucoma implant).
  Interventions: Procedure: Tube shunt surgery
- Trabeculectomy with Mitomycin C (Experimental): Participants in this group will receive a Trabeculectomy surgery with Mitomycin C
  Interventions: Procedure: Trabeculectomy; Drug: Mitomycin C

INTERVENTIONS:
Procedure: Tube shunt surgery — The procedure involves implantation of a Baerveldt consisting of a tube that is connected to an end plate. The tube is inserted into the anterior chamber and shunts aqueous humor to the end plate located in the equatorial region of the eye. The aqueous humor is then absorbed by the tissues around the eye.
  Other Names: Baerveldt glaucoma implant
  Arms: Tube shunt surgery group
Procedure: Trabeculectomy — The procedure involves removal of a small portion of trabecular meshwork and adjacent tissue under a partial thickness scleral flap. Aqueous humor drains into the subconjunctival space producing a filtering bleb. The aqueous humor then diffuse out of the bleb.
  Arms: Trabeculectomy with Mitomycin C
Drug: Mitomycin C — A fluid retaining sponge soaked in 0.4 mg/ml Mitomycin C will be applied in the region of Trabeculectomy site for about 2 minutes
  Arms: Trabeculectomy with Mitomycin C

SUMMARY:
The purpose of the Primary Tube Versus Trabeculectomy (PTVT) Study is to compare the long-term safety and efficacy of nonvalved tube shunt surgery to trabeculectomy with mitomycin C in eyes that have not had previous ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* Glaucoma that is inadequately controlled on tolerated medical therapy with Intraocular Pressure (IOP) greater than or equal to 18 mm Hg and less than or equal to 40 mm Hg
* No previous incisional ocular surgery

Exclusion Criteria:

* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits
* Pregnant or nursing women
* No light perception vision
* Active iris neovascularization or active proliferative retinopathy
* Iridocorneal endothelial syndrome
* Epithelial or fibrous ingrowth
* Chronic or recurrent uveitis
* Steroid-induced glaucoma
* Severe posterior blepharitis
* Unwilling to discontinue contact lens use after surgery
* Previous cyclodestructive procedure
* Conjunctival scarring from prior ocular trauma or cicatrizing disease precluding a superior trabeculectomy
* Functionally significant cataract
* Need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Gedde, MD, Study Chair — Bascom Palmer Eye Institute; Dale K Heuer, MD, Study Chair — Medical College of Wisconsin; Richard K Parrish, MD, Study Chair — Bascom Palmer Eye Institute
Locations (16):
- United States (12):
  - University of California Davis Medical Center, Sacramento, California
  - University of Florida, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas
  - University of Texas, Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- University of Toronto, Toronto, Canada
- United Kingdom (3):
  - Moorfields Eye Hospital, London
  - St. Thomas' Hospital, London
  - Queen Mary's Sidcup Hospital, Sidcup

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gedde SJ, Chen PP, Heuer DK, Singh K, Wright MM, Feuer WJ, Schiffman JC, Shi W; Primary Tube Versus Trabeculectomy Study Group. The Primary Tube Versus Trabeculectomy Study: Methodology of a Multicenter Randomized Clinical Trial Comparing Tube Shunt Surgery and Trabeculectomy with Mitomycin C. Ophthalmology. 2018 May;125(5):774-781. doi: 10.1016/j.ophtha.2017.10.037. Epub 2017 Dec 18. PMID 29248173
- [Result] Gedde SJ, Feuer WJ, Lim KS, Barton K, Goyal S, Ahmed IIK, Brandt JD; Primary Tube Versus Trabeculectomy Study Group. Treatment Outcomes in the Primary Tube Versus Trabeculectomy Study after 3 Years of Follow-up. Ophthalmology. 2020 Mar;127(3):333-345. doi: 10.1016/j.ophtha.2019.10.002. Epub 2019 Oct 9. PMID 31727428
- [Result] Gedde SJ, Feuer WJ, Shi W, Lim KS, Barton K, Goyal S, Ahmed IIK, Brandt J; Primary Tube Versus Trabeculectomy Study Group. Treatment Outcomes in the Primary Tube Versus Trabeculectomy Study after 1 Year of Follow-up. Ophthalmology. 2018 May;125(5):650-663. doi: 10.1016/j.ophtha.2018.02.003. Epub 2018 Feb 21. PMID 29477688
- [Result] Gedde SJ, Feuer WJ, Chen PP, Heuer DK, Singh K, Wright MM; Tube Versus Trabeculectomy and Primary Tube Versus Trabeculectomy Study Groups. Comparing Treatment Outcomes from the Tube Versus Trabeculectomy and Primary Tube Versus Trabeculectomy Studies. Ophthalmology. 2021 Feb;128(2):324-326. doi: 10.1016/j.ophtha.2020.06.059. Epub 2020 Jul 2. PMID 32622848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Started | 125 | 117
Completed | 91 | 87
Not Completed | 34 | 30
Not completed — Death | 5 | 5
Not completed — Lost to Follow-up | 29 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C | Total
Number analyzed (Participants) | 125 | 117 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.4) | 60.8 (12.3) | 61.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 84 | 76 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 59 | 57 | 116
  White | 50 | 45 | 95
  Hispanic | 9 | 6 | 15
  Asian | 6 | 7 | 13
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Failure
Description: Surgical failure is defined as:
  1. Inadequate Intraocular Pressure (IOP) Reduction (IOP > 21 mmHg or reduced < 20% below baseline on 2 consecutive follow-up visits after 3 months)
  2. Reoperation for glaucoma
  3. Persistent hypotony (IOP ≤ 5 mmHg on 2 consecutive visits after 3 months)
  4. Loss of light perception vision
Time Frame: Up to 5 years
Population: The number of participants requiring glaucoma operations includes only those that had a failed surgery due to glaucoma reoperation.
Measure: Count of Participants; unit: Participants
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
Participants
  Inadequate IOP reduction | 31 | 23
  Reoperation for Glaucoma | 18 | 9
  Loss of light perception vision | 0 | 1
  Persistent Hypotony | 0 | 5

2. Secondary Outcome: Intraocular Pressure
Description: Intraocular pressure will be reported in mmHg and measured using Goldmann applanation tonometry or a Tono-Pen.
Time Frame: At baseline, At 1 year, At 18 months, At 2 years, At 3 years, At 4 years, At 5 years
Population: Participants who underwent additional glaucoma surgery were censored from analysis after reoperation. Not all participants completed all visits to complete the IOP assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
mmHg
  Intraocular Pressure: Baseline | 23.3 (4.9) | 23.9 (5.7)
  Intraocular Pressure: 1 year: number analyzed (Participants) | 108 | 105
  Intraocular Pressure: 1 year | 13.8 (4.1) | 12.4 (4.4)
  Intraocular Pressure: 18 months: number analyzed (Participants) | 99 | 97
  Intraocular Pressure: 18 months | 13.5 (4.1) | 12.8 (4.7)
  Intraocular Pressure: 2 years: number analyzed (Participants) | 99 | 96
  Intraocular Pressure: 2 years | 13.6 (3.9) | 12.9 (5.2)
  Intraocular Pressure: 3 years: number analyzed (Participants) | 87 | 88
  Intraocular Pressure: 3 years | 13.9 (4.2) | 12.1 (4.8)
  Intraocular Pressure: 4 years: number analyzed (Participants) | 83 | 79
  Intraocular Pressure: 4 years | 13.5 (3.5) | 13.5 (5.4)
  Intraocular Pressure: 5 years: number analyzed (Participants) | 74 | 75
  Intraocular Pressure: 5 years | 13.4 (3.5) | 13.0 (5.2)

3. Secondary Outcome: Number of Participants With Reported Postoperative Complications
Description: Number of participants with early and late postoperative complications will be reported as per treating physician assessment
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
Participants
  Early Postoperative Complications | 24 | 40
  Late Postoperative Complications | 27 | 32

4. Secondary Outcome: Visual Acuity Using a Snellen Chart
Description: Visual acuity will be measured using a Snellen chart on logMAR (Logarithm of Minimal Angle of Resolution) scale. Letter-by letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: At Baseline, At 5 years
Population: Not all participants were able to complete the 5 year follow up visit and assessments.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
logMAR
  Baseline | 0.20 (0.42) | 0.25 (0.51)
  5 years: number analyzed (Participants) | 91 | 87
  5 years | 0.30 (0.54) | 0.42 (0.21)

5. Secondary Outcome: Visual Acuity as Measured Using EDTRS Chart
Description: Visual acuity will be reported as the number of correctly identified letters on the Early Treatment Diabetic Retinopathy Study (EDTRS) chart. Total score ranges from 0-100 with the higher score indicating better visual acuity.
Time Frame: At baseline, At 5 years
Population: Not all participants were able to complete the 5 year follow up visit and assessments.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
letters
  Baseline | 73 (20) | 73 (20)
  5 years: number analyzed (Participants) | 91 | 87
  5 years | 69 (23) | 66 (27)

6. Secondary Outcome: Visual Field
Description: Visual fields will be measured using standard automated perimetry.
Time Frame: Up to 5 years
Population: No data is reported for this outcome as data can not be extracted from system despite exhausting all efforts to do so.
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Reoperation for Glaucoma
Description: The number of participants requiring reoperation for glaucoma will be reported
Time Frame: Up to 5 years
Population: The number of participants requiring glaucoma operations includes those that had a failed surgery due to glaucoma reoperation, as well as, other patients who failed because of inadequate intraocular pressure reduction and subsequently underwent glaucoma surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
Participants | 21 | 12

8. Secondary Outcome: Number of Glaucoma Medications
Description: The need for supplemental glaucoma medications will be reported as the number of glaucoma medications used
Time Frame: At Baseline, At 1 year, At 18 months, At 2 years, At 3 years, At 4 years, At 5 years
Population: Participants who underwent additional glaucoma surgery were censored from analysis after reoperation. Not all participants completed all visits to complete assessment.
Measure: Mean (Standard Deviation); unit: glaucoma medications used
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
Number analyzed (Participants) | 125 | 117
glaucoma medications used
  Baseline | 3.1 (1.1) | 3.2 (1.1)
  1 year: number analyzed (Participants) | 108 | 105
  1 year | 2.1 (1.4) | 0.9 (1.4)
  18 months: number analyzed (Participants) | 99 | 97
  18 months | 2.1 (1.3) | 0.8 (1.3)
  2 years: number analyzed (Participants) | 99 | 96
  2 years | 2.2 (1.0) | 1.0 (1.5)
  3 years: number analyzed (Participants) | 87 | 88
  3 years | 2.1 (1.4) | 1.2 (1.5)
  4 years: number analyzed (Participants) | 83 | 79
  4 years | 2.3 (1.4) | 1.3 (1.4)
  5 years: number analyzed (Participants) | 74 | 75
  5 years | 2.2 (1.3) | 1.3 (1.4)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Tube Shunt Surgery Group | Trabeculectomy With Mitomycin C
All-Cause Mortality (participants affected / at risk) | 5/125 | 5/117
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/117
Other Adverse Events (participants affected / at risk) | 51/125 | 72/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tube Shunt Surgery Group (N=125) | Trabeculectomy With Mitomycin C (N=117)
Shallow or flat anterior chamber (Eye disorders) | 15 (15) | 15 (15)
Choroidal Effusion (Eye disorders) | 11 (11) | 12 (12)
Wound Leak (Surgical and medical procedures) | 1 (1) | 13 (13)
Hyphema (Eye disorders) | 8 (8) | 5 (5)
Encapsulated bleb (Eye disorders) | 13 (13) | 26 (26)
Hypotony Maculopathy (Eye disorders) | 1 (1) | 6 (6)
Wound Dehiscence (Surgical and medical procedures) | 2 (2) | 0 (0)
Aqueous Misdirection (Eye disorders) | 0 (0) | 1 (1)
Corneal Dellen (Eye disorders) | 1 (1) | 0 (0)
Cystoid Macular Edema (Eye disorders) | 3 (3) | 0 (0)
Suture-related infection (Infections and infestations) | 0 (0) | 1 (1)
Persistent Diploplia (Eye disorders) | 5 (5) | 3 (3)
Dysethesia (Eye disorders) | 1 (1) | 3 (3)
Persistent Corneal Edema (Eye disorders) | 0 (0) | 3 (3)
Iritis (Eye disorders) | 2 (2) | 1 (1)
Bleb Leak (Eye disorders) | 0 (0) | 1 (1)
Conjunctival Cyst (Eye disorders) | 1 (1) | 0 (0)
Anterior Bleb Migration with Irregular Astigmatism (Eye disorders) | 0 (0) | 1 (1)
Plate erosion (Eye disorders) | 1 (1) | 0 (0)
Tube retraction (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-05-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT00666237/Prot_SAP_ICF_000.pdf